CLINICAL TRIAL: NCT00741936
Title: Chinese Herbal Medicine for Functional Constipation: A Randomized, Double-blind, Placebo Controlled Trial
Brief Title: An Effectiveness and Safety Study of Chinese Herbal Medicine for Functional Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Food and Health Bureau, Hong Kong (Other Government); Purapharm International (Hk) Ltd. (Industry)
Responsible Party: Principal Investigator, ZhaoXiang Bian, Professor, Director of Clinical Division, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PID-002
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Results first posted 2011-12-16 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2015-03

CONDITIONS: Functional Gastrointestinal Disorders; Constipation
Keywords: Functional Constipation; Chinese Herbal Medicine; MaZiRenWan; Hemp Seed Pill; Traditional Chinese Medicine; Herbal Medicine
MeSH Terms: conditions — Gastrointestinal Diseases; Constipation | interventions — ma zi ren wan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MaZiRenWan (MZRW) (Experimental): MZRW granule, 7.5g/sachet
  Interventions: Drug: MaZiRenWan (MZRW)
- Placebo (Placebo Comparator): Placebo granule, 7.5g/sachet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MaZiRenWan (MZRW) — MZRW granule dissolved in 150ml hot water (oral), 7.5g/sachet, twice daily
  Other Names: Hemp Seed Pill
  Arms: MaZiRenWan (MZRW)
Drug: Placebo — Placebo granule dissolved in 150ml hot water (oral), 7.5g/sachet, twice daily
  Other Names: MZRW Placebo
  Arms: Placebo

SUMMARY:
Functional constipation (FC) is a common complaint in clinical practice, but treatment for this condition in conventional medicine is suboptimal. Complementary and alternative medicines, especially Chinese herbal medicine (CHM) are used frequently by patients, however, there is little research evidence about these commonly used CHM. The purpose of the study is evaluate the efficacy and safety of an ancient CHM formula, MaZiRenWan (MZRW), by comparing with placebo.

DETAILED DESCRIPTION:
Constipation is a common gastrointestinal complaint in clinical practice, which affects in estimated 12%-19% of American, 14% of Asian, and up to 27% of the population depending on demographic factor, sampling, and definition. With the unsatisfactory response to current symptomatic treatments, many patients seek help from traditional Chinese medicine (TCM), mostly by taking Chinese herbal medicine (CHM).

According to the TCM theory, constipation can be broadly divided into two types, excessive and deficient, based on the underlying aetiology. The former is characterized by the presence of Heat or pathological accumulation of Qi. Heat causes constipation by drying the Intestines and the stool. Patients present with hard, dry, pellet like stool, red complexion, dry mouth or halitosis, red tongue with a dry yellow coat, and slippery and rapid pulse. Qi stagnation causes constipation by disrupting the normal movement and descent of Stomach and Intestinal Qi. Patients present difficulty in passing stools, feelings of incomplete evacuation, abdominal distension or pain, frequent belching and flatulence, tongue with thin coat and wiry pulse. The latter, deficient constipation, is delineated as the dryness from insufficient fluid lubrication in the form of blood or lack of propulsion power from the deficiency of Qi or Yang. Besides, the treatment approaches vary from syndrome to syndrome.

The formula of MaZiRenWan (MZRW) composed of six Chinese herbs is firstly recorded in a TCM classic, Discussion of Cold-induced Disorders (Shang Han Lun), and it has been commonly used for constipation in excessive pattern throughout Asia since the Han Dynasty (A.D. 200). By combining the actions of these herbs, MZRW can moisten the Intestines, drain heat, promote the movement of Qi and unblock the bowel. Although previous studies show that MZRW has purgative and laxative effects and may be useful for functional constipation (FC), there are significant methodological weaknesses. Furthermore, the dose of CHM intervention being investigated from the first randomized controlled trial (RCT) published in 1983 is always based on the practitioner's experience, TCM literatures, or experts' comments, but not the results from stringent clinical trials, such as dose determination study. Therefore, the evidence produced will be attenuated or even misleading if improper dose is taken.

In the present study, the efficacy and safety of MZRW in optimal dosage were justified by comparing with placebo under strict clinical trial design.

ELIGIBILITY:
Inclusion Criteria:

* Meet of Rome III diagnostic criteria of functional constipation
* Meet the diagnosis of Excessive Constipation according to the TCM theory
* Age of 18 to 65 years (inclusive)
* Complete spontaneous bowel movement (CSBM)≦2times/wk
* Severity of constipation≧4pts (7 pts scale from 0 to 6pts) and the overall scoring of constipation-related symptoms≧8pts (6items in 7pts scale) for self symptom assessment in the run-in period
* Normal colonic evaluation (colonoscopy or barium enema) within 5 years
* Normal liver and renal function in blood test within 3 months

Exclusion Criteria:

* Drug-induced constipation
* Secondary causes of constipation (i.e. medical history of diabetes mellitus and thyroid disease)
* Abdominal surgery (i.e. Caesarean operation)
* Severe disease (i.e. cancer and acute present asthma)
* Allergy to CHM (i.e. G6PD deficiency)
* Pregnancy or breast-feeding
* Psychiatric or addictive disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-07; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhao-xiang Bian, PhD, Principal Investigator — Hong Kong Baptist University
Locations (1):
- Hong Kong Baptist University Mr. & Mrs. Chan Hon Yin Chinese Medicine Specialty Clinic and Good Clinical Practice Centre, Hong Kong, China

REFERENCES:
- [Result] Cheng CW, Bian ZX, Zhu LX, Wu JC, Sung JJ. Efficacy of a Chinese herbal proprietary medicine (Hemp Seed Pill) for functional constipation. Am J Gastroenterol. 2011 Jan;106(1):120-9. doi: 10.1038/ajg.2010.305. Epub 2010 Nov 2. PMID 21045817
- See also: Abstract — http://www.ncbi.nlm.nih.gov/pubmed/21045817

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All constipated patients (aged 18-65 years) who presented to the Chinese medicine clinics of the School of Chinese Medicine, Hong Kong Baptist University were referred. In total, 456 patients with constipation were screened from July 2008 to September 2009; of these 120 were randomized into MZRW or placebo group.
Pre-assignment Details: Many patients were excluded because they did not fulfill the inclusion criteria or they met the exclusion criteria. The demographic data and baseline variables of participants were comparable among groups
Groups:
- MaZiRenWan (MZRW): MZRW granule, 7.5g/sachet Patients were instructed to dissolve a sachet of granules in 150 ml of hot water; they took this solution orally twice daily for 8 weeks.
- Placebo: Placebo granule, 7.5g/sachet Patients were instructed to dissolve a sachet of granules in 150 ml of hot water; they took this solution orally twice daily for 8 weeks.
Period: Overall Study
Arm/Group | MaZiRenWan (MZRW) | Placebo
Started | 60 | 60
Completed | 51 | 52
Not Completed | 9 | 8
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 3 | 4
Not completed — Pregnancy | 0 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Lack of Efficacy | 0 | 2
Not completed — Low compliance | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MaZiRenWan (MZRW) | Placebo | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.72 (10.62) | 37.53 (11.42) | 37.13 (10.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 57 | 112
  Male | 5 | 3 | 8
Duration of constipation [Mean (Standard Deviation); unit: years] | 13.50 (9.96) | 15.25 (10.82) | 14.38 (10.39)
Bowel movement [Mean (Standard Deviation); unit: movements per week] | 2.79 (1.26) | 3.31 (1.61) | 3.05 (1.46)
Complete spontaneous bowel movement (CSBM) [Mean (Standard Deviation); unit: movements per week] — CSBM referred to the feeling that defecation led to complete passage of stool rather than partial or incomplete evacuation without the use of any laxative or enema within 24 hours.
  movements per week | 0.33 (0.66) | 0.52 (0.69) | 0.42 (0.68)
No. of days taking rescue therapy [Mean (Standard Deviation); unit: days per week] | 0.93 (0.17) | 0.84 (0.15) | 0.89 (1.24)
Severity of constipation [Mean (Standard Deviation); unit: Units on a scale] — It was a 7-point ordinal scale from 0=not at all to 6=very severe.
  Units on a scale | 4.47 (0.102) | 4.40 (0.10) | 4.43 (0.76)

OUTCOME MEASURES:

1. Secondary Outcome: Responder of Complete Spontaneous Bowel Movement (CSBM)
Description: Participants with a mean increase of complete spontaneous bowel movement (CSBM)>=1 movement per week compared with the last 14 days of the run-in period were defined as responders.
  CSBM referred to the feeling that defecation led to complete passage of stool rather than partial or incomplete evacuation without the use of any laxative or enema within 24 hours.
Time Frame: End of follow up (wk18)
Population: Statistical analysis was performed on the population being randomized and receiving allocated intervention. Missing values were imputed by the method of last observation carried forward.
Measure: Number; unit: participants
Arm/Group | MaZiRenWan (MZRW) | Placebo
Number analyzed (Participants) | 60 | 60
participants
  Responder | 18 | 9
  Non-responder | 42 | 51
Statistical Analysis 1: Comparison: MaZiRenWan (MZRW) vs Placebo; Test type: Superiority or Other; p < 0.05, Chi-squared

2. Secondary Outcome: Bowel Movement
Time Frame: Baseline(Wk1&2), Within treatment(Wk3-10) & Within follow-up(Wk11-18)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: movements per week
Arm/Group | MaZiRenWan (MZRW) | Placebo
Number analyzed (Participants) | 60 | 60
movements per week
  Baseline(Wk1&2) | 2.79 (1.26) [2.47 to 3.12] | 3.31 (1.61) [2.89 to 3.72]
  Within treatment(Wk3-10) | 4.72 (2.37) [4.11 to 5.33] | 3.73 (1.54) [3.33 to 4.13]
  Within follow-up(Wk11-18) | 3.65 (2.23) [3.08 to 4.23] | 3.61 (1.61) [3.20 to 4.03]
Statistical Analysis 1: Comparison: MaZiRenWan (MZRW) vs Placebo; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; T-Tests were implemented: 1) between two groups of each time frame; 2) between each treatment group of each time frame and its baseline

3. Secondary Outcome: Complete Spontaneous Bowel Movement (CSBM)
Time Frame: Baseline(Wk1&2), Within treatment(Wk3-10), Within follow-up(Wk11-18)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: movements per week
Arm/Group | MaZiRenWan (MZRW) | Placebo
Number analyzed (Participants) | 60 | 60
movements per week
  Baseline (Wk1&2) | 0.33 (0.66) [0.16 to 0.49] | 0.52 (0.69) [0.34 to 0.69]
  Within treatment(Wk3-10) | 1.62 (1.98) [1.11 to 2.13] | 0.72 (1.08) [0.44 to 1.00]
  Within follow-up (Wk11-18) | 1.06 (1.67) [0.62 to 1.49] | 0.75 (1.18) [0.44 to 1.05]
Statistical Analysis 1: Comparison: MaZiRenWan (MZRW) vs Placebo; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; [statistical method as in outcome 2, analysis 1]

4. Secondary Outcome: Changes on Individual Symptom Scores
Description: It was a 7-point ordinal scale from 0=not at all to 6=very severe.
Time Frame: Baseline(Wk2), Within treatment(Wk6), End of treatment(Wk10) & End of follow-up(Wk18)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MaZiRenWan (MZRW) | Placebo
Number analyzed (Participants) | 60 | 60
Units on a scale
  Severity of constipation (Baseline) | 4.47 (0.79) [4.26 to 4.67] | 4.40 (0.74) [4.21 to 4.59]
  Severity of constipation (Wk6) | 2.82 (1.52) [2.42 to 3.21] | 3.70 (1.49) [3.32 to 4.08]
  Severity of constipation (Wk10) | 2.93 (1.43) [2.57 to 3.30] | 3.47 (1.36) [3.12 to 3.82]
  Severity of constipation (Wk18) | 3.57 (1.47) [3.19 to 3.95] | 3.63 (1.39) [3.27 to 3.99]
  Sensation of straining (Baseline) | 4.20 (0.84) [3.98 to 4.42] | 3.82 (1.20) [3.51 to 4.13]
  Sensation of straining (Wk6) | 2.60 (1.43) [2.23 to 2.97] | 3.12 (1.35) [2.77 to 3.47]
  Sensation of straining (Wk10) | 2.55 (1.52) [2.16 to 2.94] | 3.28 (1.46) [2.91 to 3.66]
  Sensation of straining (Wk18) | 3.33 (1.28) [3.00 to 3.67] | 3.32 (1.37) [2.96 to 3.67]
  Incomplete of evacuation (Baseline) | 4.40 (1.12) [4.11 to 4.69] | 4.07 (1.22) [3.75 to 4.38]
  Incomplete of evacuation (Wk6) | 3.18 (1.40) [2.82 to 3.54] | 3.47 (1.49) [3.08 to 3.85]
  Incomplete of evacuation (Wk10) | 3.02 (1.51) [2.63 to 3.41] | 3.45 (1.55) [3.05 to 3.85]
  Incomplete of evacuation (Wk18) | 3.62 (1.29) [3.28 to 3.95] | 3.43 (1.57) [3.03 to 3.84]
  Sensation of bloating (Baseline) | 3.62 (1.30) [3.28 to 3.95] | 3.47 (1.33) [3.12 to 3.81]
  Sensation of bloating (Wk6) | 2.53 (1.68) [2.10 to 2.97] | 2.82 (1.76) [2.36 to 3.27]
  Sensation of bloating (Wk10) | 2.23 (1.65) [1.81 to 2.66] | 2.70 (1.81) [2.23 to 3.17]
  Sensation of bloating (Wk18) | 2.92 (1.67) [2.49 to 3.35] | 2.65 (1.83) [2.18 to 3.12]
  Sensation of abdominal pain/cramping (Baseline) | 1.98 (1.76) [1.53 to 2.44] | 1.43 (1.58) [1.03 to 1.84]
  Sensation of abdominal pain/cramping (Wk6) | 1.80 (1.60) [1.39 to 2.21] | 1.12 (1.42) [0.75 to 1.48]
  Sensation of abdominal pain/cramping (Wk10) | 1.22 (1.28) [0.89 to 1.55] | 1.07 (1.47) [0.69 to 1.45]
  Sensation of abdominal pain/cramping (Wk18) | 1.50 (1.54) [1.10 to 1.90] | 0.82 (1.35) [0.47 to 1.16]
  Sensation of nausea (Baseline) | 1.00 (1.54) [0.60 to 1.40] | 0.83 (1.45) [0.46 to 1.21]
  Sensation of nausea (Wk6) | 0.68 (1.21) [0.37 to 1.00] | 1.03 (1.57) [0.63 to 1.44]
  Sensation of nausea (Wk10) | 0.53 (0.97) [0.28 to 0.78] | 0.78 (1.30) [0.45 to 1.12]
  Sensation of nausea (Wk18) | 0.97 (1.48) [0.58 to 1.35] | 0.73 (1.53) [0.34 to 1.13]
  Passing of gas (Baseline) | 2.93 (1.75) [2.48 to 3.38] | 2.97 (1.67) [2.54 to 3.40]
  Passing of gas (Wk6) | 2.73 (1.52) [2.34 to 3.13] | 2.53 (1.70) [2.09 to 2.97]
  Passing of gas (Wk10) | 2.55 (1.43) [2.18 to 2.92] | 2.27 (1.68) [1.83 to 2.70]
  Passing of gas (Wk18) | 2.73 (1.46) [2.36 to 3.11] | 2.40 (1.60) [1.99 to 2.81]
Statistical Analysis 1: Comparison: MaZiRenWan (MZRW) vs Placebo; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; [statistical method as in outcome 2, analysis 1]

5. Secondary Outcome: Global Symptoms Improvement
Description: Participants were asked to rate their impression of change in constipation by comparing with their baseline (Wk2) at the visits during the treatment (Wk6), end of treatment (Wk10) and end of follow-up (Wk18) with scores from 0 to 6 represented markedly worse or better respectively. The response categories were collapsed to simply "improved" for score 4 to 6, "same" for score 3 or "worse" for score 0 to 2.
Time Frame: Wk 6, 10 & wk 18
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | MaZiRenWan (MZRW) | Placebo
Number analyzed (Participants) | 60 | 60
participants
  Improved (Wk6) | 49 | 28
  Same (Wk6) | 11 | 27
  Worse (Wk6) | 0 | 5
  Improved (Wk10) | 48 | 32
  Same (Wk10) | 12 | 24
  Worse (Wk10) | 0 | 4
  Improved (Wk18) | 30 | 31
  Same (Wk18) | 25 | 27
  Worse (Wk18) | 5 | 2
Statistical Analysis 1: Comparison: MaZiRenWan (MZRW) vs Placebo; Test type: Superiority or Other; p < 0.05, Chi-squared; Chi-squared test from Crosstabs analysis was implemented between two treatment groups in each time frame

6. Secondary Outcome: Success of Blinding
Description: The success of blinding was evaluated for both investigator and patients as to whether MZRW or placebo had been taken.
Time Frame: End of follow-up (Wk18)
Population: Only for subjects attended the last follow-up visit on Wk 18.
Measure: Number; unit: participants
Units Other Than Participants: No. of subjects attended last visit
Arm/Group | MaZiRenWan (MZRW) | Placebo
Number analyzed (Participants) | 60 | 60
Number analyzed (No. of subjects attended last visit) | 54 | 55
participants
  Subjects with correct guessing | 32 | 16
  Investigator with correct guessing | 42 | 27
Statistical Analysis 1: Comparison: MaZiRenWan (MZRW) vs Placebo; Test type: Superiority or Other; p = 0, simple percentage

7. Primary Outcome: Responder of Complete Spontaneous Bowel Movement (CSBM)
Description: Patients with a mean increase of ≧1 complete spontaneous bowel movement(CSBM)/wk compared with the baseline(wk1-2) will be defined as responders. CSBM referred to the feeling that defecation led to complete passage of stool rather than partial or incomplete evacuation without the use of any laxative or enema within 24 hours.
Time Frame: End of treatment (wk10)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | MaZiRenWan (MZRW) | Placebo
Number analyzed (Participants) | 60 | 60
participants
  Responder | 26 | 5
  Non-responder | 34 | 55
Statistical Analysis 1: Comparison: MaZiRenWan (MZRW) vs Placebo; Test type: Superiority or Other; p < 0.05, Chi-squared

8. Secondary Outcome: Blood Urea Level
Time Frame: Pre-treatment (Wk2) & Post-treatment (Wk10)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | MaZiRenWan (MZRW) | Placebo
Number analyzed (Participants) | 60 | 60
mmol/L
  Pre-treatment (Wk2) | 3.87 (1.03) | 3.98 (0.93)
  Post-treatment (Wk10) | 4.01 (0.97) | 4.24 (1.11)
Statistical Analysis 1: Comparison: MaZiRenWan (MZRW) vs Placebo; Test type: Superiority or Other; p < 0.05, Paired-samples t-test; Paired-Samples T Test was implemented between pre-treatment (Wk2) and post-treatment (Wk10) of each treatment group

9. Secondary Outcome: Blood Creatinine Level
Time Frame: Pre-treatment (Wk2) & Post-treatment (Wk10)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | MaZiRenWan (MZRW) | Placebo
Number analyzed (Participants) | 60 | 60
μmol/L
  Pre-treatment (Wk2) | 66.67 (9.48) | 66.05 (7.91)
  Post-treatment (Wk10) | 66.90 (9.20) | 64.62 (7.40)
Statistical Analysis 1: Comparison: MaZiRenWan (MZRW) vs Placebo; Test type: Superiority or Other; p < 0.05, Paired-Samples T Test; Paired-Samples T Test was implemented between pre-treatment (Wk2) and post-treatment (Wk10) of each treatment group

10. Secondary Outcome: Serum Glutamic Pyruvic Transaminase(SGPT) Level
Time Frame: Pre-treatment (Wk2) & Post-treatment (Wk10)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | MaZiRenWan (MZRW) | Placebo
Number analyzed (Participants) | 60 | 60
U/L
  Pre-treatment (Wk2) | 15.82 (7.81) | 14.05 (4.87)
  Post-treatment (Wk10) | 14.70 (5.50) | 13.68 (4.55)
Statistical Analysis 1: Comparison: MaZiRenWan (MZRW) vs Placebo; Test type: Superiority or Other; p < 0.05, Paired-Samples T Test; Paired-Samples T Test was implemented between pre-treatment (Wk2) and post-treatment (Wk10) of each treatment group

11. Secondary Outcome: Serum Glutamic Oxaloacetic Transaminase (SGOT)
Time Frame: Pre-treatment (Wk2) & Post-treatment (Wk10)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | MaZiRenWan (MZRW) | Placebo
Number analyzed (Participants) | 60 | 60
U/L
  Pre-treatment (Wk2) | 17.82 (4.05) | 17.77 (3.91)
  Post-treatment (Wk10) | 17.20 (3.45) | 17.12 (4.27)
Statistical Analysis 1: Comparison: MaZiRenWan (MZRW) vs Placebo; Test type: Superiority or Other; p < 0.05, Paired-Samples T Test; Paired-Samples T Test was implemented between pre-treatment (Wk2) and post-treatment (Wk10) of each treatment group

ADVERSE EVENTS:
Time Frame: Within the whole 18 weeks study period
Arm/Group | MaZiRenWan (MZRW) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 11/60 | 7/60
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MaZiRenWan (MZRW) (N=60) | Placebo (N=60)
Abdominal pain / cramping or bloating (Gastrointestinal disorders) | 8 | 2
nausea or stomach discomfort (Gastrointestinal disorders) | 4 | 4
diarrhea and passing of gas (Gastrointestinal disorders) | 1 | 0
dizziness or headache (General disorders) | 1 | 2
palpitations and trembling hands (General disorders) | 0 | 1
difficulty in micturition (Renal and urinary disorders) | 1 | 0 — Subject with a history of hyperplastic prostate
aggravation of rhinitis symptoms (General disorders) | 1 | 0 — Subject with history of rhinitis.
skin itching (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No